CLINICAL TRIAL: NCT07375108
Title: A Multi-center Quasi-experimental Study in Northern Italy to Evaluate the Impact of Sepsis Bundle in Obstetric Settings: the SOS Study
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Raffaele Bruno, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: SOS
Record Dates: First submitted 2025-12-18; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sepsis Newborn; Sepsis
MeSH Terms: conditions — Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- An initial group of women hospitalized between May 1, 2015, and May 1, 2018, before the regional doc
  Interventions: Other: microbiological results from blood cultures or other materials.
- A second group of women hospitalized from January 1, 2019, to January 1, 2022, following the introdu

INTERVENTIONS:
Other: microbiological results from blood cultures or other materials. — Data will be collected regarding outcomes, demographic and clinical characteristics of patients, as well as microbiological results from blood cultures or other materials. The information will be extracted from available electronic or paper hospital medical records.
  Groups: An initial group of women hospitalized between May 1, 2015, and May 1, 2018, before the regional doc

SUMMARY:
Despite advances in the diagnosis and treatment of sepsis, the studies available in the literature report very high maternal and fetal/neonatal mortality and morbidity in cases of sepsis occurring during pregnancy or the puerperium. It is the third leading cause of maternal death after postpartum hemorrhage and eclamptic syndrome.

Since 2002, the Surviving Sepsis Campaign (SSC) has emphasized the importance of standardized guidelines (sepsis bundles) for the management of sepsis and septic shock in the general population, with the goal of improving patient outcomes. Randomized controlled trials have not produced consistent results regarding the actual impact of sepsis bundles on reducing mortality and morbidity.

There are even fewer studies specifically addressing maternal sepsis.

In May 2018, a Regional Operational Guidance Document for the early identification and management of sepsis in obstetrics was approved and distributed (Decree No. 7691 of 28/05/2018). It contains recommendations addressed to all healthcare facilities in the Lombardy region that have Gynecology and Obstetrics services, as well as to those facilities that, although lacking such services, might still be required to manage pregnancy-related issues.

The purpose of this document is to standardize diagnostic and therapeutic procedures in order to allow early recognition and prompt management, aimed at reducing complications of sepsis in obstetrics, in accordance with the 2016 Surviving Sepsis Campaign guidelines.

Our study aims to evaluate the impact of the aforementioned regional decree on the management of maternal sepsis in the main maternity hospitals in Lombardy.

In particular, we will assess the effect of the decree and its implementation on the length of hospital stay for patients diagnosed with sepsis during pregnancy and the puerperium. Secondary objectives will also include evaluating in-hospital mortality, the number of transfers to the Intensive Care Unit, and the incidence of complications related to the septic event, such as premature rupture of membranes, preterm birth, miscarriage, and fetal or perinatal death.

We will compare two populations of women hospitalized with a diagnosis of sepsis during pregnancy or the puerperium, before and after the approval and dissemination of the regional bundle.

In parallel, we will assess the appropriateness of blood culture requests and observe the incidence of the different microorganisms responsible for the septic event.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older;
* pregnancy or postpartum;
* patient discharged with a diagnosis of sepsis reported on the Hospital Discharge Form, in accordance with the Surviving Sepsis Campaign guidelines.

Exclusion Criteria:

- no exclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: and adult patients discharged with a Hospital Discharge Form reporting the diagnosis of sepsis (or related complications) during pregnancy or the postpartum period hospitalized in the Gynecology and Obstetrics Units of five hospitals in Lombardy.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the Regional Guideline Document for the Early Identification and Management of Sepsis in Obstetrics | 1 Year
  Evaluate the effectiveness of the Regional Guideline Document for the Early Identification and Management of Sepsis in Obstetrics (Decree No. 7691 of May 28, 2018) in reducing the length of hospital stay of women admitted with a diagnosis of sepsis durin

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Malattie Infettive 1, Pavia, Pavia, Italy